CLINICAL TRIAL: NCT00185549
Title: An Interactive Program to Improve Care for Children With Cystic Fibrosis
Brief Title: An Interactive Program to Improve Care for Children With CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 78910
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-10-05 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis;; patient education,; Internet
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Behavioral: CF. DOC

SUMMARY:
The purpose of this study is to evaluate the impact of an internet based program for children and families (CF.DOC) with Cystic Fibrosis on health outcomes. The program provides for virtual visits, a personal health record, messaging with clinicians and several tools for monitoring self-care behaviors. We anticipate that this intervention will provide for more intensive monitoring and feedback of self-care behaviors and will lead to improved health status and in particular nutritional status

DETAILED DESCRIPTION:
Subjects will be drawn from the pool of children who receive their care at the LPCH/Stanford Cystic Fibrosis Center. A letter will be sent to all eligible patients inviting them to participate in the study. This letter will also be available in the CF clinic. All subjects who agree to participate in the study will have the study described to them by a research assistant either in person or over the phone. Informed consent will be obtained all on subjects. Subject who elect to participate will be randomized into either an intervention group or a control group . Subjects in the intervention group will be given Internet Access to the program CF.DOC. They will also be given training in how to use the program for communication with their clinicians, participating in a virtual visit and using online forms and surveys. Subjects in the control group will be advised that they will receive usual care and will have access to CF.DOC at the completion of the study. At the beginning of the study and at 3 month intervals subjects will be asked to complete a cystic fibrosis Quality of life survey. At the beginning and end of the study all subjects will complete a patient experience questionnaire (CAPHS 2.0 CCC supplement ) and an CF.DOC evaluation survey. As part of their regular care all subjects will also have their nutritional status measured and pulmonary function assessed. subjects in the intervention group will asked to define treatment goals that are important to them (e.g. attending camp or participating in sports) and to define health measures that will help monitor progress in meeting these goals e.g. weekly weights or pulmonary function. Subjects in the intervention group will be asked to log onto CF.DOC at least one time per month.

ELIGIBILITY:
Inclusion Criteria: Patients with Cystic Fibrosis diagnosed by a sweat chloride analysis and/or testing for the CF gene between the ages of 1 month and 21 years of age. Patients must also be English speaking -

Exclusion Criteria: Non-English speaking patients

-

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2004-03; Study Completion 2005-09

PRIMARY OUTCOMES:
Improvement in nutritional status
Improvement in CF related quality of life

SECONDARY OUTCOMES:
Phone utilization
COmponents of program liked and dis-liked

CONTACTS AND LOCATIONS:
Overall Officials: David A Bergman, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States